CLINICAL TRIAL: NCT05440604
Title: Nutrient and Immunity Status in Children Aged 3-5 Years Consuming Their Habitual Diet With or Without Fortified Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020.01.INF
Record Dates: First submitted 2022-06-27; First posted 2022-07-01 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Nutritional Status; Child Nutrition Sciences; Toddlers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fortified milk group (Experimental): 2 daily servings of the investigational fortified milk for 16 weeks
  Interventions: Other: Fortified milk
- Observational group (No Intervention): will be asked to consume beverages in accordance with their habitual pattern of intake

INTERVENTIONS:
Other: Fortified milk — Commercially available milk-based fortified beverage that has an updated profile of key micronutrients along with appropriate levels of protein and other macro- and micro- nutrients, in accordance with global and local nutritional recommendations
  Arms: Fortified milk group

SUMMARY:
This study compares the status of key micronutrients (vitamins A, C, D, E, and zinc) in young children given investigational fortified milk versus young children consuming their habitual pattern of beverage intake (milk and non-milk beverages).

DETAILED DESCRIPTION:
Hypothesis that Vitamin A, C, D, E and zinc status of children consuming 2 servings / day of fortified milk for 16 weeks will be better than those of children consuming their habitual pattern of beverage intake (milk and non-milk beverages, juices, sugar-sweetened drinks) for the same duration. This is based on previous study findings that (i) the toddler's and preschooler's diet, in reality, are often not optimal, putting toddlers and preschool age children at risk of insufficient intakes of several nutrients, and (ii) consuming fortified milk supplemented with these nutrients might provide optimal intakes of these nutrients.

ELIGIBILITY:
Inclusion Criteria:

1. Having obtained his/her parent's(s') or his/her legal guardian written informed consent and signed and dated informed consent.
2. Child's parent(s)/guardian is/are of legal age of consent, must understand the informed consent and other study documents, and is/are willing and able to fulfill the requirements of the study protocol
3. Age 3 years old to 4 years old and 6 months at enrolment
4. Healthy at birth, singleton, full-term gestational birth (37-42 completed weeks of gestation), with a birth weight of 2.5 kg to 3.9 kg
5. At the time of enrolment, the participant's weight-for-age, height-for-age, weight-for-height, BMI z-score should be within -2 to +1
6. At the time of enrolment, the participant is in good health (no history of underlying metabolic or chronic disease; congenital malformation; or any other condition which, in the opinion of the investigator, is likely to interfere with: the ability of the child to ingest food, the normal growth and development of the child, or the evaluation of the infant; acute illness in a minor condition which are common in childhood such as viral or bacterial infection e.g. conjunctivitis, otitis media, upper/lower respiratory tract infection, gastroenteritis, hand foot & mouth disease at time of enrolment is permitted) as determined by physical history, physical exam and judgement by the investigator
7. Child's parent(s)/guardian can be contacted directly by telephone or mobile phone throughout the study

Exclusion Criteria:

1. Chronic infectious, metabolic, genetic illness, or other disease including any condition that impacts feeding, or any outcome measures
2. Child exhibits any clinical signs of potential micronutrient deficiencies (e.g., hemoglobin < 100 g/L based on screening assessment, rickets based on physical exam).
3. Known or suspected cows' milk protein intolerance / lactose intolerance /allergy or severe food allergies that impact diet
4. Breast milk used exclusively / mixed in place of all other milk, and/or milk alternatives at 3 years of age
5. Consuming supplement(s) of relevance to the study outcome relating diet to status, vitamins A, D, E and C; zinc
6. Child's family who in the Investigator's judgment cannot be expected to comply with the protocol or study procedures

Ages: 36 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
change in vitamin A status | 16 weeks
  measure in serum retinol in μmol/L
change in vitamin C status | 16 weeks
  measure in plasma vitamin C in mg/dL
change in vitamin D status | 16 weeks
  measure in serum 25-hydroxy vitamin D (25[OH]D) in nmol/L
change in vitamin E status | 16 weeks
  measure in plasma alpha-tocopherol in mg/L
change in zinc status | 16 weeks
  measure in plasma zinc in μg/dl

SECONDARY OUTCOMES:
monitor growth and development | 16 weeks
  anthropometry assessment measured by weight (kg)
monitor growth and development | 16 weeks
  anthropometry assessment measured by height (cm)
monitor growth and development | 16 weeks
  anthropometry assessment measured by BMI (kg/m^2)
assess dietary intake | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  using a 24-hour Dietary Recall completed by the parent / caregiver
assess habitual pattern of food and beverage intake | 16 weeks
  using a semi-quantitative food frequency questionnaire completed by the parent / caregiver
assess child developmental milestones | 16 weeks
  using Laban Quotient to assess physical, social, self-help and cognitive; minimum score 1 , maximum 5; higher scores indicate more positive outcomes
assess fortified milk acceptability | 4 weeks, 8 weeks, 12 weeks, 16 weeks
  using Milk Intake Diary for interventional group completed by the parent / caregiver
nucleotides status assessment | 16 weeks
  measure concentration of nucleotides
monitor standard adverse events (AE) | 16 weeks
  safety assessment by monitoring the AEs linked with participation in study
monitor absenteeism from day care or pre-school due to illness | 16 weeks
  safety assessment by monitoring the days of absenteeism linked with participation in study
monitor concomitant medication (CM) reporting | 16 weeks
  safety assessment by monitoring number of participants that took concomitant medication linked with participation in study

CONTACTS AND LOCATIONS:
Overall Officials: Elvira M Estorninos, MD, Principal Investigator — Las Piñas Doctors Hospital
Locations (1):
- Las Piñas Doctors Hospital, Las Piñas, National Capital Region, Philippines